CLINICAL TRIAL: NCT02623881
Title: The Effectiveness of Cervical Pessary Versus Vaginal Progesterone for Preventing Premature Birth in IVF Twin Pregnancies: a Randomized Controlled Trial.
Brief Title: Cervical Pessary vs. Vaginal Progesterone for Preventing Premature Birth in IVF Twin Pregnancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vietnam National University (Other)
Collaborators: Mỹ Đức Hospital (Other)
Responsible Party: Principal Investigator, Manh Tuong Ho, Doctor, Vietnam National University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCKH/CGRH_10_2015
Record Dates: First submitted 2015-11-30; First posted 2015-12-08 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Pregnancy
Keywords: Cervical pessary; Vaginal progesterone; Twins; Premature birth
MeSH Terms: conditions — Premature Birth | interventions — Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cervical pessary (Active Comparator): Cervical pessary (Arabin) will be inserted to participants at 16-22 weeks and removed at 36 weeks of pregnancy or in case of premature rupture of membranes, signs of preterm labour or patient severe discomfort.
  Interventions: Device: Cervical pessary
- Vaginal Progesterone (Active Comparator): Vaginal progesterone (Cyclogest 400 mg) once a day will be used, from 16-22 to 36 weeks of pregnancy or in case of premature rupture of membranes, signs of preterm labour or patient severe discomfort.
  Interventions: Drug: Vaginal progesterone

INTERVENTIONS:
Device: Cervical pessary — Arabin (cervical pessary) will be inserted at 16-22 weeks and removed at 36 weeks of pregnancy or in case of premature rupture of membranes, signs of preterm labour or patient severe discomfort
  Other Names: Arabin
  Arms: Cervical pessary
Drug: Vaginal progesterone — Vaginal progesterone (Cyclogest 400 mg) once a day will be used, from 16-22 to 36 weeks of pregnancy or in case of premature rupture of membranes, signs of preterm labour or patient severe discomfort
  Other Names: Cyclogest 400mg
  Arms: Vaginal Progesterone

SUMMARY:
To compare the effectiveness of cervical pessary (Arabin) and vaginal progesterone for preventing premature birth in twin pregnancies after IVF

DETAILED DESCRIPTION:
This will be a randomized controlled trial.

Women with twin pregnancies, at 16-22 weeks of gestation, will be invited to participate into the study.

Subjects meeting the study criteria will be randomized into two groups: (1) treated with cervical pessary (Arabin) or (2) treated with 400mg vaginal progesterone, once daily. Randomization will be done by third party via telephone, using a computer generated random list, with a variable block size of 2, 4 or 8. Apart from randomization, patients will be examined and treated according to local protocol.

Patients in pessary group will have an Arabin pessary placed within a week after randomization. A pessary certified by European Conformity (CE0482, MED/CERT ISO 9003/ EN 46003; Dr. Arabin, Witten, Germany) will be inserted through the vagina of the woman in the recumbent position and will be placed upward around the cervix. The research-team members who inserted the Arabin pessary have experience with Arabin pessary for singleton pregnancy before.

Patients in progesterone group will use vaginal progesterone (Cyclogest 400mg) once daily before bedtime, starting from the day of randomization onwards. They will be given a monitoring sheet and instructed to note everyday the date of using. If they forget one dose of any night, and remember it in the next morning or afternoon, they will use immediately the forgotten dose and continue with the dose of that day at night. If one dose is missed until the next evening, there will be no compensation use, they will only use the dose of the next day. Any change in using medication should be noted in the monitoring sheet.

In both groups, intervention will be stopped at 36 weeks of gestation or at delivery. All the participants will have follow-up visits every 4 weeks. If patients develop (threatened) preterm labor, they will receive treatment as routine practice.

Statistical analyses will be by intention to treat. For dichotomous endpoints, we will calculate rates. These will be compared by calculating a relative risk and a 95% confidence interval. Between-group differences in non-continuous variables will be assessed using the χ2-test. Results of continuous variables were given in mean ± SD or in percentage. Between-group differences of continuous variables were assessed with the Student's t-test. We will consider correlation between neonatal endpoints when we analyse at the level of the child. We assessed time to delivery by Cox proportional hazard analysis and Kaplan-Meier estimates, and compared results with a log-rank test. We plan an exploratory subgroup analysis in women with a cervical length of less than the 25th percentile (according to the distribution in all twins), as well as 25th - 50th percentile, 50th - 75th percentile and > 75th percentile. We also plan an exploratory subgroups analyses for chorionicity. A p-value < 0.05 will be considered to indicate a statistically significant difference. The analysis will be done with statistical Package for Social Sciences version 19 (SPSS, USA).

Sample size has been set at 290. This was incorporated in an amendment of the protocol, and was approved by the IRB on 22 Sept 2016.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for enrolment into this trial, each female subject must fulfil all of the following criteria at the start of enrolment, unless specified otherwise:

* Women with a twin pregnancy (mono- and di-chorionic)
* 16 0/7 to 22 0/7 weeks of gestation
* Maternal age ≥ 18 yrs
* Cervical length less than 38 mm
* Informed consent
* Not participating in another PTB study at the same time

Exclusion Criteria:

To be eligible for enrolment in this study each subject must not meet any of the following criteria:

* History of cervical surgery
* Cervical cerclage in place
* Twin-to-twin transfusion syndrome
* Stillbirth or major congenital abnormalities in any of the fetus
* Severe vaginal discharge, acute vaginitis
* Premature rupture of membranes
* Premature labor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-03-04 (Actual); Primary Completion 2017-11-02 (Actual); Study Completion 2017-11-02 (Actual)

PRIMARY OUTCOMES:
Preterm birth before 34 weeks of gestation | At birth
  Birth before 34 weeks

SECONDARY OUTCOMES:
Intrauterine death before 24 weeks of gestation | From randomisation to 24 weeks
  Death of any fetus intrauterine before 24 weeks
Stillbirth | At birth
  Baby born with no signs of life at or after 28 weeks
Delivery before 24 weeks of gestation | At birth
  Birth before 24 weeks
Delivery before 28 weeks of gestation | At birth
  Birth before 28 weeks
Delivery before 32 weeks of gestation | At birth
  Birth before 32 weeks
Delivery before 37 weeks of gestation | At birth
  Birth before 37 weeks
Labour induction | At birth
  Labor initiated with a method such as oxytocin, Foley bulb, or artificial rupture of membranes.
Prelabour rupture of membrane | From randomization to less than 37 weeks
  Prelabour rupture of membranes and gestational age less than 37 weeks
Mode of delivery | At birth
  Spontaneous, forceps/ventouse, emergency C-section, planned C-section
Livebirth at any gestational age | At birth
  Birth of at least one newborn that exhibits any sign of life, such as respiration, heartbeat, umbilical pulsation or movement of voluntary muscles
Use of tocolytics drug | From 24 weeks to 34 weeks
  Use of tocolytics drug to prevent premature labor
Use of corticosteroids | From 24 weeks to 34 weeks
  Use of corticosteroids to prevent respiratory distressed syndrome
Admission days for preterm labor | From 24 weeks to 37 week
  Days admission to hospital due to preterm labor
Choriamnionitis | From randomization to birth
  Intraamniotic infection
Maternal morbidity | From randomization to birth
  Thromboembolic complications, urinary tract infection treated with antibiotics, pneumonia, endometritis, hypertension disorder, eclampsia or HELLP syndrome, or death
Birthweight | At birth
  Weight of babies
Birthweight < 1500g | At birth
  Weight of babies < 1500g
Birthweight < 2500g | At birth
  Weight of babies < 2500g
Congenital anomalies | At birth
  Congenital malformation of newborn
5-minute Apgar score | At birth
  Apgar score at 5 minute after birth
5-minute Apgar score < 7 | At birth
  Apgar score < 7 at 5 minute after birth
Admission to NICU | Within 7 days after delivery
  The admittance of newborn to NICU
Length of NICU admission | Up to 28 days after birth
  Number of days admittance of newborn to NICU
Severe respiratory distress syndrome | Within 24 hours after delivery
  Grade 2 or worse, as diagnosed by Giedion et al
Bronchopulmonary dysplasia | At time of discharge home or at 36 weeks of gestational age
  Diagnosed according to the international consensus guideline as described by Jobe and Bancalari
Intraventricular haemorrhage | Up to 28 days after birth
  Grade II B or worse, as diagnosed by repeated neonatal cranial ultrasound by the neonatologist according to the guidelines on neuro-imaging described by de Vries et al. and Ment et al
Necrotising enterocolitis | Up to 28 days after birth
  > stage 1, will be diagnosed according to Bell
Proven sepsis | Up to 28 days after birth
  The combination of clinical signs and positive blood cultures.
Death before discharge | Up to 28 days after birth
  Death of newborn before discharge from nursery
Maternal side effects | From randomisation to birth
  Vaginal discharge, fever, other signs of infections, pain, pessary repositioning and necrosis or rupture of the cervix
Withdrawal from treatment | From randomization to 36 weeks of gestation
  Patient's discontinuation of arabin or vaginal progesterone use

CONTACTS AND LOCATIONS:
Overall Officials: Tuong M Ho, MD, Study Director — Research Center for Genetics and Reproductive Health
Locations (1):
- My Duc Hospital, Ho Chi Minh City, Tan Binh District, Vietnam

REFERENCES:
- [Derived] Dang VQ, Nguyen LK, Pham TD, He YTN, Vu KN, Phan MTN, Le TQ, Le CH, Vuong LN, Mol BW. Pessary Compared With Vaginal Progesterone for the Prevention of Preterm Birth in Women With Twin Pregnancies and Cervical Length Less Than 38 mm: A Randomized Controlled Trial. Obstet Gynecol. 2019 Mar;133(3):459-467. doi: 10.1097/AOG.0000000000003136. PMID 30741812